CLINICAL TRIAL: NCT01233713
Title: Hartmann's Versus Primary Anastomosis in Left-sided Colon Perforation - A Prospective Randomized Multicenter Trial
Brief Title: Hartmann's Versus Primary Anastomosis in Left-sided Colon Perforation
Acronym: ColonPerfRCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Winterthur KSW (Other); University of Lausanne (Other); Kantonsspital Graubünden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Colon_Perf_RCT
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Surgery; Diverticulitis; Neoplasms; Postoperative Complications
Keywords: Emergency Surgery; Bowel perforation; Diverticulitis; Neoplasms; Postoperative Complications; Randomized Controlled Trial
MeSH Terms: conditions — Diverticulitis; Neoplasms; Postoperative Complications; Intestinal Perforation | interventions — Colectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary anastomosis (Active Comparator): Primary anastomosis refers to a colonic resection with primary anastomosis and covering ileostomy, followed by a stoma reversal operation.
  Interventions: Procedure: Primary anastomosis
- Hartmann's operation (Active Comparator): Hartmann's operation is the surgical resection of the rectosigmoid colon with closure of the rectal stump and end colostomy, followed by a stoma reversal operation.
  Interventions: Procedure: Hartmann's operation

INTERVENTIONS:
Procedure: Hartmann's operation — Hartmann's operation is the surgical resection of the rectosigmoid colon with closure of the rectal stump and end colostomy, followed by a stoma reversal operation.
  Other Names: Colectomy with a proximal-end colostomy
  Arms: Hartmann's operation
Procedure: Primary anastomosis — Primary anastomosis refers to a colonic resection with primary anastomosis and covering proximal ileostomy, followed by a stoma reversal operation.
  Other Names: Colectomy, primary anastomosis and defunctioning ileostomy
  Arms: Primary anastomosis

SUMMARY:
The purpose of this multi-center randomized trial is to identify any differences in the complication rates of patients undergoing Hartmann's (end colostomy) versus Primary Anastomosis (with defunctioning ileostomy) for left-sided colonic performation (including the stoma reversal operation).

DETAILED DESCRIPTION:
Hartmann's operation: the surgical resection of the rectosigmoid colon with closure of the rectal stump and end colostomy.

End colostomy: A stoma is created from one end of the bowel while the other portion of the bowel is either removed or sewn shut (Hartmann's pouch).

The second operation (reversal) requires a colo-rectal anastomosis.

Primary anastomosis: colonic resection with primary anastomosis and defunctioning ileostomy. The second operation (stoma reversal) requires an entero-enteral anastomosis.

Anastomosis: is to join together two bowel ends to restore continuity after resection or stoma formation.

Colostomy: is a reversible surgical procedure in which a stoma is formed by drawing the healthy end of the colon through an incision in the anterior abdominal wall and suturing it into place. This opening, in conjunction with the attached stoma appliance, provides an alternative channel for feces to leave the body.

Ileostomy is a surgical opening constructed by bringing the loop of small intestine (the ileum) out onto the surface of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years
* Left-sided colon perforation
* German language speakers

Exclusion Criteria:

* Patient age < 18 years
* Perforation outside of the left-colon
* Bowel obstruction/disease without perforation
* Evidence of metastasis

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Overall post-operative complication rate defined according to the Clavien-Dindo Classification | 2006 - 2010
  The Clavien-Dindo Classification of Surgical Complications:
  Grade I: Any deviation from the normal postoperative course without the need for treatment. Grade II: Requiring pharmacological treatment with drugs. Grade III: Requiring surgical, endoscopic or radiological intervention. Grade IV: Life-threatening complication requiring IC/ICU-management. Grade V: Death of a patient

SECONDARY OUTCOMES:
Serious post-operative complication rate (Clavien-Dindo grade ≥III) for the primary operation | 2006 - 2010
  Primary operation: the one the patients were randomized to, either Hartmann's or Primary anastomosis
Serious post-operative complication rate (Clavien-Dindo grade ≥III) for the reversal operation | 2006 - 2010
  Reversal operation is the one of either the colostomy (Hartmann's) or the ileostomy (Primary anastomosis)
Overall total number of complications | 2006 - 2010
  Sum of the number of different complications
Number of complications for the primary operation | 2006 - 2010
  Primary operation is the one patients were randomized into.
Number of complications for the reversal operation | 2006 - 2010
  As above
Reversal rate | 2006 - 2010
  Reversal rate is the proportion of patients having their stoma reversed (second operation)
Operation time | 2006 - 2010
  Duration of the primary procedure, the reversal procedure, and overall (minutes)
Length of Intensive Care Unit (ICU) stay | 2006 - 2010
  In days
Length of hospital stay | 2006 - 2010
  In days
In-hospital costs | 2006 - 2010
  Cost of the primary operation, the reversal, and combined, in US dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, MD, Principal Investigator — University Hospital Zurich, Department of Visceral and Transplant Surgery, Zurich, Switzerland
Locations (4):
- Switzerland (4):
  - University Hospital Zurich, Department of Visceral and Transplant Surgery, Swiss Hepato-Pancreato-Biliary (HPB) Center, Zurich, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - University Hospital Vaudois (CHUV), Department of Visceral Surgery, Lausanne, Lausanne
  - Kantonsspital Winterthur, Winterthur, Winterthur

REFERENCES:
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Derived] Oberkofler CE, Rickenbacher A, Raptis DA, Lehmann K, Villiger P, Buchli C, Grieder F, Gelpke H, Decurtins M, Tempia-Caliera AA, Demartines N, Hahnloser D, Clavien PA, Breitenstein S. A multicenter randomized clinical trial of primary anastomosis or Hartmann's procedure for perforated left colonic diverticulitis with purulent or fecal peritonitis. Ann Surg. 2012 Nov;256(5):819-26; discussion 826-7. doi: 10.1097/SLA.0b013e31827324ba. PMID 23095627